CLINICAL TRIAL: NCT03530631
Title: Neuroimaging the Expectancy Versus Pharmacotherapy Effect of Adderall on Cognitive Performance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Karen Cropsey, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB-300000343
Record Dates: First submitted 2018-04-24; First posted 2018-05-21 (Actual); Results first posted 2019-10-14 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Expectancy Versus Pharmacotherapy Effect of Adderall
MeSH Terms: interventions — Adderall

STUDY DESIGN:
Intervention Model Description: 2 X 2, within-subjects, balanced placebo design
Who Masked: Participant, Investigator
Masking Description: This will be a double-blind study. Research assistants will administer capsules, and based on package labeling, tell the participant if they are being administered Adderall or placebo. However, researchers and participants will be blind to which medication is actually being administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Adderall/Truth (Experimental): Participants will be told they are receiving Adderall and will actually be administered Adderall.
  Interventions: Drug: Adderall
- Placebo/Truth (Placebo Comparator): Participants will be told they are receiving placebo and will actually be administered placebo.
  Interventions: Drug: Placebo
- Adderall/Deception (Experimental): Participants will be told they are receiving Adderall and will actually be administered placebo.
  Interventions: Drug: Placebo
- Placebo/Deception (Experimental): Participants will be told they are receiving placebo and will actually be administered Adderall.
  Interventions: Drug: Adderall

INTERVENTIONS:
Drug: Adderall — Participants will be administered Adderall
  Arms: Adderall/Truth; Placebo/Deception
Drug: Placebo — Participants will be administered placebo
  Arms: Adderall/Deception; Placebo/Truth

SUMMARY:
The purpose of this balanced-placebo design study is to pilot a larger study to further explore the current evidence that stimulant medications are not cognitive enhancers, despite this rampant belief in young adults. While the lack of cognitive enhancement from stimulant medication has been documented in prior research, this study is the first to utilize neuroimaging technology to examine brain regions activated during neurocognitive tasks when participants believe they have been administered stimulant medication or placebo.

DETAILED DESCRIPTION:
This is a 2 X 2 within subjects, balanced placebo design and all participants will experience each of the four conditions during four sequential weeks. Medication administered (Adderall vs. placebo) is crossed with instructional set (truth vs. deception) and participants' performance on neurocognitive tasks is compared across these groups. For example, participants are either given stimulant medication or placebo, and are either accurately told or inaccurately told that they received stimulant medication or placebo. Neuroimaging is being utilized to investigate whether participants' expectations regarding the benefits of stimulant medication affects their performance on neurocognitive tasks. The hypothesis of the study is that participants' expectations regarding stimulant medication will affect their performance on neurocognitive tasks, rather than the actual effect of the medication.

ELIGIBILITY:
Inclusion Criteria:

* Age (18-24)
* College student with at least average IQ
* Willingness to standardize caffeine intake to 100 mg on day of study

Exclusion Criteria:

* Attention Deficit/Hyperactivity Disorder (ADHD)
* First degree relative with ADHD
* Unwillingness to comply with caffeine specifications
* Regular use of Adderall
* Pregnant/breastfeeding
* History of substance use disorders
* Illicit stimulant use within the last year
* Contraindications to stimulants (i.e., tics, Tourette's, cardiac disease, hypertension)
* Uncontrolled medical illness
* Active contagious infection

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2018-11-10 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Cropsey, Psy.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only four subjects were recruited for this pilot study
Groups:
- Adderall Within Subjects Design: This is a within-subjects design in which participants will complete all four periods/conditions. For two sessions, participants will be accurately told that they are receiving Adderall or placebo, respectively. For two sessions, participants will be inaccurately informed that they are receiving Adderall or placebo. The participants will be counterbalanced across conditions to control for order effects.
Period: Adderall/Truth
Arm/Group | Adderall Within Subjects Design
Started | 4
Completed | 4
Not Completed | 0
Period: Placebo/Truth
Arm/Group | Adderall Within Subjects Design
Started | 4
Completed | 4
Not Completed | 0
Period: Adderall/Deception
Arm/Group | Adderall Within Subjects Design
Started | 4
Completed | 4
Not Completed | 0
Period: Placebo/Deception
Arm/Group | Adderall Within Subjects Design
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Adderall Within Subjects Design
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Consistently Attending and Completing Four Neuroimaging Sessions
Description: Using a balanced placebo design, participants were either administered mixed amphetamine salts or placebo. Their cognitive performance was assessed in the MRI scanner. The main outcome measure was the feasibility of participants attending four neuroimaging sessions.
Time Frame: A total of 4 imagining sessions, an average of 60 minutes each
Measure: Count of Participants; unit: Participants
Arm/Group | Adderall/Truth | Placebo/Truth | Adderall/Deception | Placebo/Deception
Number analyzed (Participants) | 4 | 4 | 4 | 4
Participants | 4 | 4 | 4 | 4

ADVERSE EVENTS:
Time Frame: Baseline to one month
Arm/Group | Adderall/Truth | Placebo/Truth | Adderall/Deception | Placebo/Deception
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT03530631/Prot_001.pdf